CLINICAL TRIAL: NCT03459326
Title: Sexuality of the Man Whose Couple is Taken Care of in Medical Assistance to Procreation. Study of Case Witnesses
Acronym: AMPlaisir
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-383; 2017-A00902-51 (Other: 2017-A00902-51)
Record Dates: First submitted 2018-03-02; First posted 2018-03-08 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Men in Relation; Couple Whose Taken Care in Medical Assisted to Reproduction
Keywords: male sexuality; medical assisted to procreation; International Index of Erectile Function questionnaire

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- control group: men in relation
  Interventions: Other: IIEF (International Index of Erectile Function questionnaire )
- FIV group: men whose couple taken care of fecundation in vitro
  Interventions: Other: IIEF (International Index of Erectile Function questionnaire )
- ICSI group: men whose couple taken care of intracytoplasmic injection
  Interventions: Other: IIEF (International Index of Erectile Function questionnaire )
- IUI group: men whose couple taken care of intrauterine insemination
  Interventions: Other: IIEF (International Index of Erectile Function questionnaire )

INTERVENTIONS:
Other: IIEF (International Index of Erectile Function questionnaire ) — The questionnaire is presented and answered without help. Answers to the IIEF Questionnaire will be collected in order to obtain the following scores (the total score is of no interest):
  * Erectile function (score 1 to 30)
  * Orgasmic function (score 0 to 10)
  * Desire (score 2 to 10)
  * Sexual satisfaction (score 0 to 15)
  * Overall satisfaction (score 2 to 10)

SUMMARY:
According to the World Health Organization and the World Association for Sexual Health, sexual health is directly associated with the psychological well-being and quality of life of each individual.

Infertility is a real public health problem. In recent years, there has been a clear decline in male fertility in industrialized countries, particularly in sperm quality. Male infertility may be perceived as a loss of masculinity and so men will be more reluctant to talk about their fertility problem than women. The studies published so far have focused on infertile men without any specification on the type or stage of care in Medically assisted procreation (MAP).

Through our work, we propose to evaluate the impact of the type of care in Medical Assistance with procreation on the sexuality of man. Does the type of MAP technique used (intrauterine insemination, in vitro fertilization or intra cytoplasmic sperm injection) have an impact on male sexuality? Sexual health and reproductive health are closely linked; management of sexual disorders is essential to improve the quality of life. A prevention of sexual difficulties during the care of these patients in MAP can be set up in the MAP service from Clermont-Ferrand hospital.

The main objective of our study is therefore to evaluate the perceived quality of sexuality by the man whose couple is engaged in a process of medical assistance to procreation.

DETAILED DESCRIPTION:
Infertility is a real public health problem. In recent years, there has been a clear decline in male fertility in industrialized countries, particularly sperm quality. In the general population, 70% of desired pregnancies are obtained after 6 months and 90% after one year of unprotected intercourse. A couple is considered infertile in the absence of pregnancy after one year of unprotected sex. Currently about 15% of couples of childbearing age is 1 in 7 couples consult for infertility. A French team evaluated the infertility etiologies. Among 1686 couples, infertility was female in 33% of cases, male in 20% of cases and mixed in 39% of cases. Infertility was said to be unexplained in 8% of the couples evaluated.

Male partners of infertile couples experience significantly higher stress and sexual dysfunction during the fertile period compared to the non-fertile period. The high stress levels are probably due to the psychological pressure associated with efforts to conceive but certainly also with the forced moment of sexual intercourse around the ovulatory cycle of the partner. Sexuality can therefore be deprived of its recreational and erotic value and subordinated to the purpose of pregnancy. The man and the woman become "spawners" and the love relationship is organized towards a procreative goal, affecting the spontaneity of the relationship of the couple. Sexual intercourse then proceeds less and less from erotic desire and more and more desire for pregnancy. The man who doubts his fertility is ready to adjust his sexuality for greater efficiency in order to obtain the child, which represents his personal reassurance and the social proof of his sexual power. Sexual desire disorders are therefore the most frequent sexual disorder in infertile couples. Treatments and medical requirements to treat infertility may be responsible for inhibiting sexual desire. Indeed, sex becomes impersonal and driven by medical procedures. Medical assistance with procreation (MAP) is becoming increasingly important in our society. In 2011 according to the figures of the agency of biomedicine, 23 127 children were born thanks to the attempts of MPAs made, or 2.8% of children born in the general population that same year. However, MAP techniques do not always lead to pregnancy, according to the figures of the weekly epidemiological bulletin on 100 couples who start IVF:

* 41 will have a child thanks to IVF
* 59 will not have them in the context of IVF:

  * 7 will have a child with another treatment
  * 11 will have a child naturally
  * 11 will adopt a child
  * 30 couples will not have children

Infertile men may feel stigmatized because they are perceived to be deficient in a specific component of their masculinity. When men discover their infertility, men usually go through a crisis. This crisis represents a manifestation of long-standing anxiety about the nature of man, his role and function. The confusion of fertility, power and masculinity has consequences for infertile men. Male infertility can be perceived as a loss of masculinity. Men will be more reluctant to talk about their fertility problem than women. The literature suggests that the exams and the vocabulary of consultation also contribute to the anxiety of loss of male sexual identity, of self-deprecation in men. The diagnosis announcement is an important moment of care. This announcement should be cautious and the words cleverly chosen because the narcissistic injury can be profound. The team of Marci et al evaluated the impact of the diagnosis of infertility on sexuality. It could be shown that men newly diagnosed as infertile presented lower scores compared to fertile controls. This team showed that during the early stages of the diagnosis of infertility, the sexual life of couples was reached. An observational study also showed that 11% of the men had failed in the second collection because of a diagnosis of infertility. Patients in the fertile group had inferior spermatic characteristics compared with patients in the fertile group without significant difference. In the literature, a higher prevalence of erectile dysfunction in infertile men is reported compared to the general male population. The team of Khademi in 2008 show that 61.8% of patients have sexual dysfunction including 2% with severe erectile dysfunction. An observational study evaluated a total of 1,468 infertile men and 942 fertile men. The incidences of premature ejaculation (PE) and erectile dysfunction (ED) in the infertile group were significantly higher than those in the fertile group (PE: 19.01% vs. 10.93%, P <0.001; ED: 18.05% vs. 8.28%, P <0.001). In addition, anxiety and depression were more prevalent among infertile men compared to fertile men (anxiety: 38.01% vs 26.65%, p <0.001, depression: 15.74% vs. 10.08% P <0.001). Some authors reported that sexual arousal was maintained during the management of infertility. Other results have reported a decrease in sexual arousal. Despite the difficult stages they are going through, the 2 partners treated for infertility maintain a good understanding within their couple and support each other. The studies published so far have focused on infertile men without any specification on the type or stage of management of MPA. Similarly, the type of infertility encountered is rarely mentioned. Only one study assessed concordance between sperm characteristics and sexual dysfunction.

The main objective of our study is therefore to evaluate the perceived sexual quality by the man whose couple is cared for in MAP. It is an exploratory study of the control case type. This work will make it possible to evaluate the impact of the type of treatment in MAP on the sexuality of the man. Does the techniques used in MAP (Intra uterine insemination, in vitro fertilization or intra cytoplasmic sperm injection) have an impact on male sexuality? In order to be able to quantify sexual dysfunction in this study, the IIEF: the international index of erectile function questionnaire will be given to the included patients. The IIEF is an internationally validated test and translated in several languages. This questionnaire has been the subject of several publications especially in the field of infertility (Bechoua et al., 2016). It allows to assign a score of erectile dysfunction (severe score 1 to 10, moderate score 11 to 16, low to moderate score 17 to 21, low score 22 at 25, no erectile dysfunction score 26 to 30). This test also classifies sexual dysfunction under several domains.

Erectile function: item 1, 2, 3, 4, 5 and 15 (score 1 to 30) Orgasmic function: item 9 and 10 (score 0 to 10) Desire: item 11 and 12 (score 2 to 10) Sexual satisfaction: items 6, 7 and 8 (score 0 to 15) Overall satisfaction: item 13 and 14 (score 2 to 10)

Men are often left behind and may be disinvested from MAP protocols. Depending on the results, patients who have a significant impact on their sexuality of their care in MAP can be diagnosed and supported with the establishment of a sexology consultation in the service. Conducting a study of this type in the MAP service from CHU Estaing in Clermont-Ferrand will open a space of expression complementary.

ELIGIBILITY:
Inclusion Criteria:

* for witnesses : men in relation
* for cases : men in relation and whose couple taken care of medical assisted to procreation (IUI, FIV, ICSI)

Exclusion Criteria:

* for witnesses : single men
* for cases : men whose couple supported with gamete donation
* Men with viral risk

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men in relation
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2017-11-07 (Actual); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Perception of sexual quality by man | at day 1
  In order to quantify sexual dysfunction, the International Index of Erectile Function questionnaire (IIEF) will be given to patients included. The IIEF is an internationally validated test. It is used to assign a score of erectile dysfunction: severe score 1 to 10; moderate score 11 to 16; low to moderate score 17 to 21; Low score 22 to 25; no erectile dysfunction score 26 to 30

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie MESTRES, MD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France